CLINICAL TRIAL: NCT00867464
Title: Extended Follow-Up of Young Women in Costa Rica Who Received Vaccination Against Human Papillomavirus Types 16 and 18 and Unvaccinated Controls
Brief Title: Extended Follow Up of Young Women in Costa Rica Who Received Vaccine for Human Papillomavirus Types 16 and 18 and Unvaccinated Controls
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCI-2016-00231; NCI-2016-00231 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 999909106; 09-C-N106 (Other: National Cancer Institute)
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-07

CONDITIONS: Anal Carcinoma; Cervical Carcinoma; Human Papillomavirus Infection; Human Papillomavirus-Related Cervical Carcinoma; Oral Cavity Carcinoma
MeSH Terms: conditions — Anus Neoplasms; Uterine Cervical Neoplasms; Papillomavirus Infections; Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (long term follow-up): Participants undergo long term follow-up comprising risk factor questionnaire, pelvic examination for all sexually experienced women, and specimen collection at years 6, 8, and 10.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Other: Long-term Follow-up; Other: Questionnaire Administration

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Correlative studies
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Long-term Follow-up — Undergo extended follow-up
  Other Names: long term follow-up (clinical study); long-term follow-up (research); LTFU
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial studies extended follow up of young women in Costa Rica who received vaccine for human papillomavirus types 16 and 18 and unvaccinated controls. Collecting information from young women in Costa Rica who have received vaccine for human papillomavirus types 16 and 18 and a new group of unvaccinated controls enrolled for the follow-up period, may help doctors learn more about the risks and benefits of prophylactic human papillomavirus vaccine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the 10-year global impact of human papillomavirus (HPV)-16/18 vaccination of young adult women.

II. To evaluate determinants of the immune response to HPV and the vaccine, and markers of long-term protection.

III. To evaluate the natural history of HPV and cervical disease in vaccinated and unvaccinated populations.

OUTLINE:

Participants undergo long term follow-up comprising risk factor questionnaire, pelvic examination for all sexually experienced women, and specimen collection at years 6, 8, and 10.

ELIGIBILITY:
Inclusion Criteria:

* Women who participated in the Costa Rica Vaccine Trial (CVT) and lived in the Guanacaste province and a few areas of Puntarenas closest to Guanacaste will be eligible for the long-term follow up LTFU study
* Women who received the HPV-16/18 vaccine at the start of CVT will be invited for up to 6 years of additional follow-up, and women who were originally in the control arm of CVT and were offered the HPV-16/18 vaccine at crossover will be invited for an additional 2 years of follow-up
* A subset of the control arm women who are in the crossover immunogenicity subcohort will be followed the full 6 years
* Some women who received HPV vaccination and were not invited into the LTFU protocol (stopped attending their screening visits during CVT, discontinued their study participation during CVT or lived outside the study area) will be invited to participate in the LTFU protocol, particularly those who received an incomplete vaccination schedule
* UNVACCINATED CONTROL GROUP:
* Born in or between July 1978 and November 1987
* Residents of Guanacaste Province and a few areas of Puntarenas closest to Guanacaste at some point during 2005
* Able to speak/understand Spanish
* Apparently mentally competent
* Written informed consent obtained prior to enrollment

Exclusion Criteria:

* History of cervical cancer
* History of hysterectomy
* Any important medical condition or other criteria that the investigator considers that precludes enrollment
* Vaccination with Gardasil or Cervarix will be an exclusionary criterion, but few women are expected to have received these vaccines at the time of enrollment; use of these vaccines after enrollment is not a criterion for study interruption but we plan to collect information on vaccination history so that the few women who report having been vaccinated with one of the HPV vaccines after enrollment can be evaluated separately at analysis

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Young women in Costa Rica who received vaccination against human papillomavirus types 16 and 18 and unvaccinated controls.
Sampling Method: Non-Probability Sample
Enrollment: 8670 (Estimated)
Dates: Start 2009-03-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative rate of cervical intraepithelial neoplasia 3 (CIN3) | At 10 years
  Both absolute rate differences and percent reduction in rates will be evaluated.
Level of immune response markers as prediction of long-term success of HPV vaccine | Up to 10 years
  For efficiency, a nested case-control approach is envisioned to evaluate this question. We propose to compare women who become infected against a subset of those who do not (non-failures) with respect to immune response markers of interest.
Increase in the rate of cervical lesions associated with other carcinogenic HPV types that the vaccine does not protect against from prevention of HPV-16/18 associated cervical lesions through vaccination | Up to 10 years
  The 10-year cumulative rate of incident CIN2+ associated with HPV types other than HPV-16/18 and closely related HPV types in the alpha-7/9 species for which evidence of vaccine cross-protection is demonstrated will be compared between vaccinated and unvaccinated women.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Kreimer, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Agencia Costarricense de Investigaciones Biomédicas (ACIB), Liberia, Guanacaste Province, Costa Rica

REFERENCES:
- [Derived] Shing JZ, Hu S, Herrero R, Hildesheim A, Porras C, Sampson JN, Schussler J, Schiller JT, Lowy DR, Sierra MS, Carvajal L, Kreimer AR; Costa Rica HPV Vaccine Trial Group. Precancerous cervical lesions caused by non-vaccine-preventable HPV types after vaccination with the bivalent AS04-adjuvanted HPV vaccine: an analysis of the long-term follow-up study from the randomised Costa Rica HPV Vaccine Trial. Lancet Oncol. 2022 Jul;23(7):940-949. doi: 10.1016/S1470-2045(22)00291-1. Epub 2022 Jun 13. PMID 35709811
- [Derived] Porras C, Tsang SH, Herrero R, Guillen D, Darragh TM, Stoler MH, Hildesheim A, Wagner S, Boland J, Lowy DR, Schiller JT, Schiffman M, Schussler J, Gail MH, Quint W, Ocampo R, Morales J, Rodriguez AC, Hu S, Sampson JN, Kreimer AR; Costa Rica Vaccine Trial Group. Efficacy of the bivalent HPV vaccine against HPV 16/18-associated precancer: long-term follow-up results from the Costa Rica Vaccine Trial. Lancet Oncol. 2020 Dec;21(12):1643-1652. doi: 10.1016/S1470-2045(20)30524-6. PMID 33271093